CLINICAL TRIAL: NCT00882856
Title: Treating Clozapine-induced Sinustachycardia With Bisoprolol - a Double Blinded Placebo Controlled Cross Over Study
Brief Title: Treating Clozapine-induced Sinustachycardia With Bisoprolol
Acronym: Biscloz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-09215-22/5.1. 22AUG2011
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Clozapine-induced Sinustachycardia
Keywords: Clozapine; Sinustachycardia; Heartrate variability; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bisoprolol-washout -placebo (Active Comparator): Bisoprolol - wash out - placebo
  Interventions: Drug: Bisoprolol; Drug: Placebo
- Placebo - wash out - bisoprolol (Active Comparator): Placebo - wash out - bisoprolol
  Interventions: Drug: Bisoprolol; Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol "Vitabalnas" 10 mg once daily
  Other Names: Bisoprolol "Vitabalans"
Drug: Placebo — placebo

SUMMARY:
Clozapine-induced sinustachycardia occurs in 25% of patients treated with clozapine and sustained sinustachycardia might be a risk factor for dilated cardiomyopathy. This double-blinded cross over placebo controlled study investigate whether 10 mg bisoprolol are efficient in treating clozapine-induced sinustachycardia measured as heart rate, heart rate variability, QTc and T-wave morphology.

ELIGIBILITY:
Inclusion Criteria:

* Treated with clozapine > 3 months and minimum 100 mg/day
* Fixed dose 14 days before inclusion
* Heart rate > 100 (ECG)
* Pregnancy test negative
* Clozapine-induced sinustachycardia documented by ECG or case record
* Sexual abstinence or contraception
* Informed consent

Exclusion Criteria:

* Substance abuse
* Physical diseases, contraindications for clozapine or bisoprolol
* Asthma or chronic obstructive lung disease
* Blood pressure < 100/60 or recent history of syncopes
* QTc>500 ms, SA-block, AV- block II or III
* Restrictions by Danish mental act
* Allergic to clozapine or bisoprolol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | Baseline, visit 1+2+3

SECONDARY OUTCOMES:
QTc, T-wave morphology and other ECG markers | Baseline, visit 1+2+3
Hamilton-Anxiety scale | Baseline, visit 1+2+3
Salivation rate | Baseline, visit 1+2+3
Orthostatic blood pressure | Baseline, visit 1+2+3
WHO-QoL | Baseline, visit 1+2+3
Nocturnal Hypersalivation Rating Scale (NHRS). | Baseline, visit 1+2+3

CONTACTS AND LOCATIONS:
Overall Officials: Ole Schjerning, M.D., Study Director — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Psychiatry, Aalborg, Denmark